CLINICAL TRIAL: NCT05587205
Title: Phase 1, Randomized, Masked, Sham-Controlled Study to Assess the Safety and Tolerability of EO2002 in Subjects Undergoing Cataract Surgery
Brief Title: Safety and Tolerability of EO2002
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Collaborators: Emmecell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: VSH-002
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Cataract; Endothelial Cell Loss, Corneal
MeSH Terms: conditions — Cataract; Corneal Endothelial Cell Loss | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: 2 arms are masked as indicated and 2 arms are open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment at time of surgery (Experimental): EO2002 intracameral injection
  Interventions: Biological: EO2002
- Treatment post surgery (Experimental): EO2002 intracameral injection
  Interventions: Biological: EO2002
- Treatment at time of or post surgery (Active Comparator): EO2002 intracameral injection
  Interventions: Biological: EO2002
- Sham injection at time of or post surgery (Sham Comparator): Sham injection
  Interventions: Other: Sham injection

INTERVENTIONS:
Biological: EO2002 — Intracameral injection of a single dose of magnetic human corneal endothelial cells (EO2002) either at the time of cataract surgery or post-cataract surgery
  Other Names: Magnetic Human Corneal Endothelial Cells
  Arms: Treatment at time of or post surgery; Treatment at time of surgery; Treatment post surgery
Other: Sham injection — Sham injection
  Arms: Sham injection at time of or post surgery

SUMMARY:
The goal of this clinical study is to assess the safety of intracameral injection of EO2002 in subjects post-cataract surgery.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years.
2. Subject has uncomplicated history of cataract that has progressed to a level requiring standard cataract extraction with intraocular lens implant surgery.
3. Decreased endothelial cell count

Exclusion Criteria:

All ocular criteria apply to study eye unless otherwise noted.

1. Other corneal disease
2. Macular disease that in the investigator and/or sponsor's opinion would limit the ability of the subject to demonstrate improvement in BCVA.
3. Descemet membrane detachment.
4. History of uveitis or other ocular inflammatory disease.
5. History of incisional glaucoma surgery
6. Prior incisional eye surgery within 3 months prior to study treatment or penetrating or endothelial keratoplasty.
7. History of ocular neoplasm.
8. ETDRS BCVA in the fellow eye is worse than 35 letters (Snellen equivalent of 20/200).
9. Female who is pregnant, nursing, or planning to become pregnant, or who is of childbearing potential and not using a reliable means of contraception during the study.
10. Subject is currently participating in or has participated within the last 3 months in any other clinical trial of an investigational drug by ocular or systemic administration.
11. Any concomitant medical or psychological condition that could interfere with study participation or is otherwise not suitable for entry into the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-10-06 (Estimated); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of EO2002 | 26 weeks
  Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Endothelial Cell Density | 26 weeks
  Changes in ECD compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Sanchez Huerta, MD, Principal Investigator — Asociacion para Evitar la Ceguera
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No